CLINICAL TRIAL: NCT04936646
Title: Randomized Double-blind Study of RTMS Analgesic Effect in Chronic Neuropathic Pain. Comparison Between Three Groups: Motor Cortex Stimulation by the Classic Coil B65, Deeper Stimulation by the Coil B70 and Placebo Stimulation. Analysis of Long-term RTMS-induced Brain Changes Using FMRI.
Brief Title: Study of RTMS Analgesic Effect in Chronic Neuropathic Pain,
Acronym: NEUROSTIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 38RC20192
Record Dates: First submitted 2021-06-03; First posted 2021-06-23 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Chronic Neuropathic Pain
Keywords: rTMS; Chronic neuropathic pain; Repetitive Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Classic rTMS Stimulation using the B65 Coil (Experimental)
  Interventions: Device: RepetitiveTranscranial Magnetic Stimulation (rTMS)
- Deeper rTMS Stimulation using the B70 Coil (Experimental)
  Interventions: Device: RepetitiveTranscranial Magnetic Stimulation (rTMS)
- control group with a sham stimulation using a sham coil (Sham Comparator)
  Interventions: Device: RepetitiveTranscranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: RepetitiveTranscranial Magnetic Stimulation (rTMS) — The rTMS protocol consist of one session per day for five days during the first week, then three sessions the second week and then one session the third week, followed by two monthly sessions.

SUMMARY:
The purpose of this study is to compare the analgesic effectiveness of three modes of repetitive Transcranial Magnetic Stimulation (rTMS) in chronic neuropathic pain:

* Classical rTMS stimulation
* Deeper rTMS stimulation
* Sham rTMS stimulation

DETAILED DESCRIPTION:
Conduct of study:

* Entry into the study: After informed consent, patients will be randomised. The physician responsible for conducting neurostimulation sessions will make the randomization via an interactive web response system (IWRS). Only this physician will have the knowledge of the group allocated to the patient.
* Baseline : Patients, will record on a diary form, a daily Visual Numeric Scale(VNS) of Pain Intensity for 1 week.
* Treatment sessions: after the baseline, sessions of neurostimulation will begin for seven weeks.
* After the end of neurostimulation sessions, patients will be followed for 2 weeks.
* Throughout their participation in the study, patients will plot on a diary form their daily VNS.

ELIGIBILITY:
Inclusion Criteria:

* Patient's written consent
* Affiliated with social security system
* Male or female, suffering for more than a year from unilateral refractory neuropathic pain: hemi-body, upper limb, lower limb and facial chronic pain.
* Patient whose analgesic treatment, is stable for at least 1 month.
* Patient not responding to conventional treatments
* Prescreening EVN >3

Exclusion Criteria:

* History of drug addiction, epilepsy, cranial trauma
* History of psychiatric disorder
* Patients previously treated with rTMS
* Patient with intracranial ferromagnetic material or implanted stimulator
* New treatment for less than one month
* Pregnant or Breastfeeding woman
* Patient who does not understand the study protocol
* Persons who are protected under the act.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-07-16 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Evolution of Pain. | Pain progression will be assessed from week 1 (before treatment) to week 7 (end of treatment)
  Comparison between the 3 groups of the evolution of the weekly value of the Visual Numeric Scale (VNS): The patient will raise his pain level on a follow-up diary each day. The VNS average will be calculated for each week. The NSV is a 10-point scale, ranging from 0 (worse) to 10 (better).

SECONDARY OUTCOMES:
Assesment of Potential Changes in Sensory-motor Cortical Maps Induced by rTMS | Day 60 from the beginning of rTMS treatment compared to baseline.
  Comparison between the 3 groups of changes in sensory-motor cortical maps using Functional magnetic resonance imaging (FMRI).
Rate of Responding Patients. | week 7 compared with baseline
  Comparison between the 3 groups of the rate of responding patients. Responding patients is defined by a 30% reduction in pain intensity assessed with VNS.
Assessment of Overall Patient Improvement. | Day 30 and day 60 from the beginning of rTMS treatment compared to baseline
  Comparison between the 3 groups of the overall patient improvement using the Clinical Global Impression of Change scale (CGI).The CGI is a 7-point scale, ranging from 1 (better) to 7 (worse).
Quality of Life Improvement. | Day 30 and day 60 from the beginning of rTMS treatment compared to baseline
  Comparison between the 3 groups of the improvement of quality of life using the SF12 (Short Form 12) questionnaire.SF12 includes a mental and social score ranging from 5.89 to 71.97 and a physical score ranging from 9.95 to 70. a high score indicates a better quality of life.
Evolution of Anxiety and Depressive Traits. | Day 30 and day 60 from the beginning of rTMS treatment compared to baseline
  Comparison between the 3 groups of the improvement of anxiety and depressive traits using the HADS questionnaire (Hospital Anxiety and Depression Scale).the HADS score varies between 0 and 42. zero corresponding to the best score.
Evolution of Symptomatological Profiles of Neuropathic Pain. | Day 30 and day 60 from the beginning of rTMS treatment compared to baseline.
  Comparison between the 3 groups of symptomatological profiles of neuropathic pain using NPSI questionnaire (Neuropathic Pain Symptom Inventory).
Sympathetic Autonomic System Injury and Small Fiber Neuropathy. | Day 60 from the beginning of rTMS treatment compared to baseline.
  Comparison between the 3 groups of sympathetic autonomic system injury and small fiber neuropathy using the Sudoscan® device.
Autonomous System Assessement. | Day 60 from the beginning of rTMS treatment compared to baseline.
  Comparison between the 3 groups of changes in skin tension and conductance during fMRI examination.
Evolution of the use of analgesic treatments. | From baseline to day 60.
  Comparison between the 3 groups of the evolution of the use of analgesic treatments reported on the diary.
Analgesic Response Analysis | From baseline to day 60.
  Comparison between the 3 groups of the evolution of the weekly EVN average according to the clinical profile of patients
Improvement of pain triggered by a stimulus (allodynia). | Day 30 and day 60 from the beginning of rTMS treatment compared to baseline.
  Comparison between the 3 groups of allodynia improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Hasan HODAJ, MD, Principal Investigator — CHUGA
Locations (1):
- Centre de la douleur, CHU Grenoble Alpes, Grenoble, Isère, France

IPD SHARING:
Plan to Share IPD: No